CLINICAL TRIAL: NCT02977715
Title: An Open-Label Prospective Cohort Study of JYNNEOS Smallpox Vaccine in Adult Healthcare Personnel at Risk for Mpox in the Democratic Republic of the Congo
Brief Title: JYNNEOS Smallpox Vaccine in Adult Healthcare Personnel at Risk for Mpox in the Democratic Republic of the Congo
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Ministry of Public Health, Democratic Republic of the Congo (Other Government); Kinshasa School of Public Health (Other); Bavarian Nordic (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: CDC-IRB-6859
Record Dates: First submitted 2016-09-07; First posted 2016-11-30 (Estimated); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Monkeypox Virus Infection
Keywords: Democratic Republic of the Congo; Modified Vaccinia Ankara (MVA); Monkeypox; Orthopoxvirus; Vaccine; Vaccinia virus; JYNNEOS; Mpox
MeSH Terms: conditions — Mpox, Monkeypox; Vaccinia | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Intervention (Liquid Formulation) (Experimental): Up to 1000 male and female healthcare personnel ages 18 years and older in Tshuapa Province in The Democratic Republic of Congo at risk for mpox will receive two doses of attenuated live virus smallpox vaccine (JYNNEOS liquid formulation) administered on days 0 and 28 via subcutaneous injection (deltoid) (1 x 10^8 Tissue Culture Infectious Dose 50 [TCID50] per 0.5 mL). A subset of participants will receive a booster dose.
  Interventions: Biological: JYNNEOS (Liquid Formulation)
- Intervention (Lyophilized Formulation) (Experimental): Up to 600 male and female healthcare personnel ages 18 years and older in Tshuapa Province in The Democratic Republic of Congo at risk for mpox will receive two doses of attenuated live virus smallpox vaccine (JYNNEOS lyophilized formulation) administered on days 0 and 28 via subcutaneous injection (deltoid) (1 x 10^8 Tissue Culture Infectious Dose 50 [TCID50] per 0.5 mL). A subset of participants will receive a booster dose.
  Interventions: Biological: JYNNEOS (Lyophilized Formulation)
- Single booster dose (Liquid Formulation) (Experimental): Up to 400 male and female healthcare personnel ages 18 years and older who received primary vaccination as a previous study participant
  Interventions: Biological: JYNNEOS (Liquid Formulation)

INTERVENTIONS:
Biological: JYNNEOS (Liquid Formulation) — Two doses of attenuated live virus smallpox vaccine (JYNNEOS liquid formulation) administered on days 0 and 28 via subcutaneous injection (deltoid) (1 x 10^8 Tissue Culture Infectious Dose 50 [TCID50] per 0.5 mL). A subset of participants will receive a booster dose.
  Other Names: Modified Vaccinia Ankara (MVA); MVA-BN; IMVAMUNE; IMVANEX
  Arms: Intervention (Liquid Formulation); Single booster dose (Liquid Formulation)
Biological: JYNNEOS (Lyophilized Formulation) — Two doses of attenuated live virus smallpox vaccine (JYNNEOS lyophilized formulation) administered on days 0 and 28 via subcutaneous injection (deltoid) (1 x 10^8 Tissue Culture Infectious Dose 50 [TCID50] per 0.5 mL). A subset of participants will receive a booster dose.
  Other Names: Modified Vaccinia Ankara (MVA); MVA-BN; IMVAMUNE; IMVANEX
  Arms: Intervention (Lyophilized Formulation)

SUMMARY:
Mpox is a febrile rash illness caused by the monkeypox virus. Its natural occurrence in the DRC puts healthcare and frontline workers at high risk of acquiring monkeypox virus infections that can prevent them from performing work duties, compromise the overall healthcare delivery in an already fragile system, and can result in death (case fatality estimates are approximately 10%).

This is an open-label prospective cohort study in up to 1,600 eligible healthcare workers at risk of mpox infection through their daily work. The study will document mpox exposure and infection in participants while concurrently evaluating the immunogenicity and safety of the vaccine, JYNNEOS (also known as MVA-BN, IMVAMUNE®, IMVANEX), in healthcare personnel in the DRC. Participation in the study is voluntary and open to male and female healthcare personnel ages 18 years and older in Tshuapa Province in The Democratic Republic of Congo who are at risk of monkeypox virus infection through their daily work or laboratory personnel performing diagnostic testing for monkeypox virus.

DETAILED DESCRIPTION:
Orthopoxvirus infections produce antibody responses that are cross-protective against other viruses within the genus. It is this property of orthopoxviruses that allows a vaccine for vaccinia virus against smallpox to be used to provide protection against mpox. Studies performed during and in the immediate aftermath of smallpox eradication demonstrated that smallpox vaccination (with a first generation vaccine) could confer protection against infection with monkeypox virus. Newer, third generation vaccines such as JYNNEOS, an attenuated (replication deficient) strain of vaccinia virus may offer an alternative safer source of vaccine-derived protection.

The clinical presentation of mpox infection is similar to smallpox, although it is less transmissible human-to-human than smallpox and less deadly (case fatality estimates for mpox are approximately 10%). Naturally-occurring human mpox is largely restricted to remote regions of the Congo Basin forest in Central Africa. This study is the first rigorous evaluation of JYNNEOS in a region where natural Orthopoxvirus transmission occurs at appreciable and predictable rates. Healthcare and frontline workers in the DRC are currently at high risk of acquiring monkeypox virus infection that prevents them from performing work duties, compromises healthcare delivery in an already fragile system, and can result in death.

This open-label prospective cohort study in up to 1,600 healthcare personnel at risk of mpox infection through their daily work will document monkeypox virus exposure and infection in vaccinated participants while concurrently evaluating the immunogenicity and safety of JYNNEOS vaccine. Study participation is voluntary and open to male and female healthcare personnel ages 18 years and older in Tshuapa Province in the DRC. Participants will receive two subcutaneous doses of JYNNEOS vaccine on days 0 and 28. A subset of study participants will receive a booster dose. Blood samples will be obtained on days 0, 14, 28, 42, 180, 365, 545, and 730 following primary vaccination for immunogenicity analysis. For individuals who receive a booster dose, blood samples will be obtained on Days 3, 7, 14, and > 1 year following booster vaccination. After each vaccination participants will be observed for at least thirty minutes. They will maintain an adverse event diary to record systemic and local adverse events for 7 days after each immunization. They will also record exposure to the monkeypox virus in an exposure diary that is reviewed at each follow-up visit.

The study will evaluate the proportion of participants who after being vaccinated 1) develop suspected or confirmed mpox infection, and 2) experience exposure to monkeypox virus. The study will also evaluate the safety and immunogenicity of JYNNEOS.

ELIGIBILITY:
Inclusion Criteria:

1. Males and nonpregnant females (as indicated by a negative urine pregnancy test prior to first dose of vaccine) age 18 years and older.
2. Healthcare personnel at risk of mpox infection working in the Tshuapa Province of DRC or laboratory personnel performing diagnostic testing for mpox at the time of enrollment
3. Willing to adhere to infection control recommendations to the extent possible based on availability of resources.
4. Able and willing to complete the informed consent process and study procedures (including blood sample collection, urine pregnancy test, and completion of adverse event diary and exposure forms).
5. Available for all study visits.

Exclusion Criteria:

1. Any history of allergy or anaphylaxis to any prior vaccines, eggs, or aminoglycosides.
2. Current pregnancy (a negative urine pregnancy test is required for women participants who self-report as not pregnant). Enrollment for such participants may be deferred to a later time at which this criteria can be met.
3. Acute illness that is accompanied by an axillary temperature ≥37.2°C (99.0°F) at the time of vaccination. Enrollment for such participants may be deferred to a later time at which this criteria can be met.
4. Known experimental research agents or other vaccine within 28 days (4 weeks) prior to vaccination. Enrollment for such participants may be deferred to a later time at which this criteria can be met.
5. Any reason the PIs suspect that data collected from this person would be incomplete or of poor quality.
6. Any condition that the PIs suspect may place the participant at an unacceptable risk of injury or render the participant unable to meet the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1600 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Monkeypox virus infection | 2 years following initial vaccination
  Proportion of participants who develop suspected or confirmed monkeypox virus infection following receipt of JYNNEOS
Monkeypox virus exposure | 2 years following initial vaccination
  Proportion of participants who experience exposure to monkeypox virus following receipt of JYNNEOS
Orthopoxvirus Antibody Response | Days 0, 14, 28, 42, 180, 365, 545, and 730 days after the receipt of the first dose of vaccine; Days 3, 7, and/or 14, and through study completion (an average of 1 year) after receipt of single booster dose of vaccine.
  Proportion of participants who have orthopoxvirus antibody responses
Distribution of Geometric Means Titers (GMTs) | Days 0, 14, 28, 42, 180, 365, 545, and 730 days after the receipt of the first dose of vaccine; Days 3, 7, and/or 14, and through study completion (an average of 1 year) after receipt of single booster dose of vaccine.
  Distribution of geometric means titers (GMTs)
Adverse event and serious adverse event information | 2 years following initial vaccination; Day 3, 7, and/or 14 after receipt of single booster dose of vaccine
  Number of participants with reported local or systemic vaccine-associated adverse events by dose, including Serious Adverse Events and Deaths

CONTACTS AND LOCATIONS:
Overall Officials: Andrea McCollum, PhD, MS, Principal Investigator — Centers for Disease Control and Prevention; Kinkodi Didine Kaba, MD, PhD, Principal Investigator — DRC
Locations (1):
- Tshuapa site, Boende, Tshuapa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petersen BW, Kabamba J, McCollum AM, Lushima RS, Wemakoy EO, Muyembe Tamfum JJ, Nguete B, Hughes CM, Monroe BP, Reynolds MG. Vaccinating against monkeypox in the Democratic Republic of the Congo. Antiviral Res. 2019 Feb;162:171-177. doi: 10.1016/j.antiviral.2018.11.004. Epub 2018 Nov 14. PMID 30445121
- [Derived] Hatmal MM, Al-Hatamleh MAI, Olaimat AN, Ahmad S, Hasan H, Ahmad Suhaimi NA, Albakri KA, Abedalbaset Alzyoud A, Kadir R, Mohamud R. Comprehensive literature review of monkeypox. Emerg Microbes Infect. 2022 Dec;11(1):2600-2631. doi: 10.1080/22221751.2022.2132882. PMID 36263798